CLINICAL TRIAL: NCT00872560
Title: Insulin Leakage and Pain Perception in IDDM Children or Adolescents, Where the Injections Are Performed With NovoFine™ 6 x 0.30 mm Needles and NovoFine® 8 x 0.30 mm Needles: An Open, Randomized, Two-period Cross-over, Multi-centre, Phase IIIb Trial at 4 Centres
Brief Title: Comparison of 2 NovoFine® Needles on the Reflux of Insulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEEDLEN/DCD/4/I
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NovoFine® needle 6 mm
  Other Names: NEEDLEN
Device: NovoFine® needle 8 mm
  Other Names: NEEDLEN

SUMMARY:
This trial is conducted in Europe. This trial aims to ensure that there is no substantial clinically relevant difference between the two Novo Nordisk needles NovoFine® 6 x 0.30 mm and NovoFine® 8 x 0.30 mm on reflux of insulin back to the surface of cutis.

ELIGIBILITY:
Inclusion Criteria:

* Children/adolescents with type 1 diabetes mellitus
* Usage of NovoPen® 1.5 for at least 3 months
* Duration of insulin treatment more than 1 year
* Normal weight according to Tanner scales
* The means of the last 2 HbA1c measurements taken within the last 6 months must be less than 10.5%

Exclusion Criteria:

* Pregnancy or desire to become pregnant
* Clinical relevant peripheral neuropathy as judged by the investigators
* Pronounced lipodystrophy in accordance with investigator's evaluation
* Use of drugs that can influence the trial
* Coagulation disorders (use of anti-coagulants)
* Serious, chronic diseases, making it highly unlikely that the subject can complete the trial

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 1998-01-20 (Actual); Primary Completion 1998-07-27 (Actual); Study Completion 1998-07-27 (Actual)

PRIMARY OUTCOMES:
Weighing of reflux of insulin | 6 seconds after injection

SECONDARY OUTCOMES:
Pain perception | after 6 weeks of treatment
Number and severity of bleedings | after 6 weeks of treatment
Reactions at injection sites | after 6 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Chieti, Italy

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com